CLINICAL TRIAL: NCT03828981
Title: A Fast-track Versus Conventional Recovery Protocol in Laparoscopic Hysterctomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Päivi Päkarinen, MD PhD Specialist on gynecologic oncology,senior consultant, gynecologic onkology, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unique Protocol ID: 98/13/03/0
Record Dates: First submitted 2019-01-21; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Gynecologic Surgery

STUDY DESIGN:
Intervention Model Description: randomized superiority trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fast-track recovery program (Active Comparator): Pre-operative Verbal and video information Tobacco cessation Daily physical activity Light meal 6 hours and clear liquids up to 2 hours before surgery No bowel preparation A warm blanket Premedication paracetamol 1g and tematsepam 20mg
  Intraoperatively For nausea and voimiting dexamethasone 10mg, dehydrobensperidol 1mg and ondancetron 4mg before emergence Analgesia: ropivacain at port sites before incision and at vaginal vault Opioids intravenously at discretion of anesthesiologist supplemented with Dexketoprofen 50mg Urinary catheter early removal Postoperative Pain: tramadol 50mg and ketoprofen100mg i.v., oral opioid if needed; patients with normal pain control receive oral pregabalin 25mg every 8 hours, paracetamol 1000mg every 8 hours, ibuprofen 600mg every 8 hours until discharge Out of bed after 2 hours from the end of surgery A liquid diet, if tolerated regular normal diet. For emesis ondansetron 4mg
  Interventions: Procedure: fast-track recovery program
- conventional recovery program (No Intervention): Preoperative preparation Verbal and written information Cessation of oral intake after previous midnight. Premedication paracetamol 1g+ diatsepam 5mg.
  Intraoperative A warm blanket at the start of procedure. Prophylaxis for nausea and vomiting: Dexamethasone 5mg at induction, and Dehydrobenzperidol 1mg, ondancetron 4mg before emergence. Analgesia: injection of ropivacain 5% 20ml at port sites at the end of surgery, Opioids i.v. (oxycodone)
  Postoperative Pain medication:Opioids i.v. (oxycodone), paracetamol 1000mg every 8 hours, ibuprofen 600mg every 8 hours Urinary catheter removal on next morning. Prolonged bowel and bed rest and gradual reintroduction of feeding.

INTERVENTIONS:
Procedure: fast-track recovery program — Pre-operative: fast-track management counseling, fast-track educational video,tobacco cessation, daily physical activity, light meal 6 hours and clear liquids up to 2 hours before surgery, no bowel preparation, a warm blanket, medication.
  Intra-operative: vaginal wound infiltrative anesthesia, early remove of urine catheter.
  Post-operative: early oral intake liquids and food, early mobilization, avoiding opioids by use of pregabaline for postoperative pain.
  Arms: fast-track recovery program

SUMMARY:
Factors affecting to length of hospital stay after fast-track recovery program in laparoscopic hysterectomy compared to conventional recovery program

DETAILED DESCRIPTION:
Factors affecting to length of hospital stay after laparoscopic hysterectomy in fast-track recovery program group compared to conventional recovery group.

The pimary outcome is time to discharge from the end of operation to discharge.

The second outcomes are amount of opioid used and NSAID, postoperative paine, nousea and vomiting, patients satisfaction, anxiety and stress-coping test, operative bleeding, operative time, postoperative complications, the cost of the laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* uterine size less than uterine size at 14 weeks of pregnancy
* at list one friend or family available to care to care after discharge.

Exclusion criteria:

* endometriosis
* contraindications to any of medications used in the study (oxycodone, ketoprofen, or paracetamol)
* language difficulties (inability to understand and speak Finnish or Swedish)
* age older that 70 years
* mental health disability that limit autonomy

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
length of hospitalisation | up to one week
  time from end of operation until discharge

SECONDARY OUTCOMES:
postoperative pain score | change in 24 hours after surgery
  Visual analog score (VAS) for pain. The scale is from 0 to 10. 0 is no pain and 10 is worst imaginable pain.
nausea | change in 24 hours after surgery
  Visual analog score (VAS) for nausea. the scale is from 0 to 10. 0 is no nausea and 10 is worst imaginable nausea.
vomiting | change in 24 hours after surgery
  Visual analog score (VAS) for vomiting. The scale is from 0 to 10. 0 is no vomiting and 10 is worst imaginable vomiting´.
complications | Up to one week.
  Frequency of complications.Values are given as n (%) and eventual complications are spesified.
The use of anelgesics for posoperative pain. | change in 24 hours after surgery
  Postoperative pain defined as total amount (mg) of analgesics used. Amount of use oxycodone (mg).
Patient quality of life | 1 month before the surgery, in the morning of surgery day and one month after surgery
  Measurement quality of life by questionnaire 15D
Patient subjective psychological stress level by general health questionnaire(GHQ12) | 1 month before the surgery, in the morning of surgery day and one month after surgery
  Measurement of psychological stress
patient quality of life | 1 month before the surgery, in the morning of surgery day and one month after surgery
  Measurement quality of life by questionnaires WHOQO-BREF

CONTACTS AND LOCATIONS:
Overall Officials: Olga Kilpiö, MD, Study Director — Helsinki University Central Hospital
Locations (1):
- Päivi Pakarinen, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No
no plan to share a data

REFERENCES:
- [Background] Borendal Wodlin N, Nilsson L, Carlsson P, Kjolhede P. Cost-effectiveness of general anesthesia vs spinal anesthesia in fast-track abdominal benign hysterectomy. Am J Obstet Gynecol. 2011 Oct;205(4):326.e1-7. doi: 10.1016/j.ajog.2011.05.043. Epub 2011 Jun 7. PMID 22083055
- [Background] Kjolhede P, Borendal Wodlin N, Nilsson L, Fredrikson M, Wijma K. Impact of stress coping capacity on recovery from abdominal hysterectomy in a fast-track programme: a prospective longitudinal study. BJOG. 2012 Jul;119(8):998-1006; discussion 1006-7. doi: 10.1111/j.1471-0528.2012.03342.x. Epub 2012 May 9. PMID 22568450
- [Background] Kjolhede P, Langstrom P, Nilsson P, Wodlin NB, Nilsson L. The impact of quality of sleep on recovery from fast-track abdominal hysterectomy. J Clin Sleep Med. 2012 Aug 15;8(4):395-402. doi: 10.5664/jcsm.2032. PMID 22893770
- [Background] Nilsson L, Wodlin NB, Kjolhede P. Risk factors for postoperative complications after fast-track abdominal hysterectomy. Aust N Z J Obstet Gynaecol. 2012 Apr;52(2):113-20. doi: 10.1111/j.1479-828X.2011.01395.x. Epub 2012 Jan 8. PMID 22224504
- [Background] Wodlin NB, Nilsson L. The development of fast-track principles in gynecological surgery. Acta Obstet Gynecol Scand. 2013 Jan;92(1):17-27. doi: 10.1111/j.1600-0412.2012.01525.x. Epub 2012 Nov 1. PMID 22880948
- [Background] Wodlin NB, Nilsson L, Kjolhede P. [Fast track has its advantages in elective gynecological surgery]. Lakartidningen. 2014 Jun 17-Jul 1;111(25-26):1120-3. No abstract available. Swedish. PMID 25072075
- [Background] Wodlin NB, Nilsson L, Kjolhede P. Health-related quality of life and postoperative recovery in fast-track hysterectomy. Acta Obstet Gynecol Scand. 2011 Apr;90(4):362-8. doi: 10.1111/j.1600-0412.2010.01058.x. Epub 2011 Feb 18. PMID 21306322
- [Background] Veenhof AA, Vlug MS, van der Pas MH, Sietses C, van der Peet DL, de Lange-de Klerk ES, Bonjer HJ, Bemelman WA, Cuesta MA. Surgical stress response and postoperative immune function after laparoscopy or open surgery with fast track or standard perioperative care: a randomized trial. Ann Surg. 2012 Feb;255(2):216-21. doi: 10.1097/SLA.0b013e31824336e2. PMID 22241289
- [Background] Wijk L, Franzen K, Ljungqvist O, Nilsson K. Implementing a structured Enhanced Recovery After Surgery (ERAS) protocol reduces length of stay after abdominal hysterectomy. Acta Obstet Gynecol Scand. 2014 Aug;93(8):749-56. doi: 10.1111/aogs.12423. Epub 2014 Jun 13. PMID 24828471
- [Background] van Bree SH, Vlug MS, Bemelman WA, Hollmann MW, Ubbink DT, Zwinderman AH, de Jonge WJ, Snoek SA, Bolhuis K, van der Zanden E, The FO, Bennink RJ, Boeckxstaens GE. Faster recovery of gastrointestinal transit after laparoscopy and fast-track care in patients undergoing colonic surgery. Gastroenterology. 2011 Sep;141(3):872-880.e1-4. doi: 10.1053/j.gastro.2011.05.034. Epub 2011 May 26. PMID 21699777
- [Background] Vlug MS, Wind J, Hollmann MW, Ubbink DT, Cense HA, Engel AF, Gerhards MF, van Wagensveld BA, van der Zaag ES, van Geloven AA, Sprangers MA, Cuesta MA, Bemelman WA; LAFA study group. Laparoscopy in combination with fast track multimodal management is the best perioperative strategy in patients undergoing colonic surgery: a randomized clinical trial (LAFA-study). Ann Surg. 2011 Dec;254(6):868-75. doi: 10.1097/SLA.0b013e31821fd1ce. PMID 21597360
- [Background] Relph S, Bell A, Sivashanmugarajan V, Munro K, Chigwidden K, Lloyd S, Fakokunde A, Yoong W. Cost effectiveness of enhanced recovery after surgery programme for vaginal hysterectomy: a comparison of pre and post-implementation expenditures. Int J Health Plann Manage. 2014 Oct-Dec;29(4):399-406. doi: 10.1002/hpm.2182. Epub 2013 May 10. PMID 23661616
- [Background] Rhou YJ, Pather S, Loadsman JA, Campbell N, Philp S, Carter J. Direct hospital costs of total laparoscopic hysterectomy compared with fast-track open hysterectomy at a tertiary hospital: a retrospective case-controlled study. Aust N Z J Obstet Gynaecol. 2015 Dec;55(6):584-7. doi: 10.1111/ajo.12093. Epub 2013 May 2. PMID 23634987
- [Background] Minig L, Chuang L, Patrono MG, Fernandez-Chereguini M, Cardenas-Rebollo JM, Biffi R. Clinical outcomes after fast-track care in women undergoing laparoscopic hysterectomy. Int J Gynaecol Obstet. 2015 Dec;131(3):301-4. doi: 10.1016/j.ijgo.2015.06.034. Epub 2015 Sep 8. PMID 26386495
- [Background] Feroci F, Lenzi E, Baraghini M, Garzi A, Vannucchi A, Cantafio S, Scatizzi M. Fast-track surgery in real life: how patient factors influence outcomes and compliance with an enhanced recovery clinical pathway after colorectal surgery. Surg Laparosc Endosc Percutan Tech. 2013 Jun;23(3):259-65. doi: 10.1097/SLE.0b013e31828ba16f. PMID 23751989
- [Background] Gouvas N, Tan E, Windsor A, Xynos E, Tekkis PP. Fast-track vs standard care in colorectal surgery: a meta-analysis update. Int J Colorectal Dis. 2009 Oct;24(10):1119-31. doi: 10.1007/s00384-009-0703-5. Epub 2009 May 5. PMID 19415308
- [Background] Hansen CT, Sorensen M, Moller C, Ottesen B, Kehlet H. Effect of laxatives on gastrointestinal functional recovery in fast-track hysterectomy: a double-blind, placebo-controlled randomized study. Am J Obstet Gynecol. 2007 Apr;196(4):311.e1-7. doi: 10.1016/j.ajog.2006.10.902. PMID 17403400
- [Background] Moller C, Kehlet H, Friland SG, Schouenborg LO, Lund C, Ottesen B. Fast track hysterectomy. Eur J Obstet Gynecol Reprod Biol. 2001 Sep;98(1):18-22. doi: 10.1016/s0301-2115(01)00342-6. PMID 11516794
- [Derived] Kilpio O, Harkki PSM, Mentula MJ, Pakarinen PI. Health-related Quality of Life after Laparoscopic Hysterectomy following Enhanced Recovery after Surgery Protocol or a Conventional Recovery Protocol. J Minim Invasive Gynecol. 2021 Sep;28(9):1650-1655. doi: 10.1016/j.jmig.2021.02.008. Epub 2021 Feb 11. PMID 33582379
- [Derived] Kilpio O, Harkki PSM, Mentula MJ, Vaananen A, Pakarinen PI. Recovery after enhanced versus conventional care laparoscopic hysterectomy performed in the afternoon: A randomized controlled trial. Int J Gynaecol Obstet. 2020 Dec;151(3):392-398. doi: 10.1002/ijgo.13382. Epub 2020 Oct 19. PMID 32961589